CLINICAL TRIAL: NCT03871296
Title: DNA Methylation in Allogeneic Hematopoietic Stem Cell Transplantation (MET_SCT_2018).
Brief Title: DNA Methylation in Allogeneic Hematopoietic Stem Cell Transplantation.
Acronym: MET_SCT_2018
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Mariarosaria Sessa, MD (Unknown); Mario Arpinati, MD (Unknown); Francesco Barbato, MD (Unknown)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 151/2018/Sper/AOUBo
Record Dates: First submitted 2019-02-04; First posted 2019-03-12 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Aging; Stem Cell Transplant Complications
Keywords: DNA-methylation; Allogeneic stem cell transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood Urine Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As a consequence of the impending increase in life expectancy, there is urgent need to adopt life-saving interventions, such as hematopoietic stem cell transplantation, (SCT) in groups of patients that have been regarded as unsuitable for such medical procedures owing to their advanced age. However, a growing body of evidence shows that age per se does not account for a reliable estimation of the capability of an individual to cope with the stressful procedure of SCT and to deal with the cognate adverse effects. Recent literature shows that changes in epigenetic markers (i.e. the extent of methylation) at specific loci of genomic DNA marks the rate of aging and allows for the estimation of the so called "biologic aging." In other words, individuals of the same chronologic age may turn out to be older or younger respect when their biologic age is assessed. This latter is expected to be tightly linked to changes in major homeostatic mechanisms and consequently to be in relationship the chance of successful SCT. The primary objective of the study is the study of DNA in patients undergoing allogeneic haematopoietic stem cell transplantation. DNA will be assessed for the extent of methylation, which will be also in relationship with circulating exogenous DNA (i.e the microbiome).

DETAILED DESCRIPTION:
The use of hematopoietic stem cell transplantation (SCT) in groups of patients previously unsuitable because of age is progressively increasing. Nowadays, allogeneic SCT in patients aged over 60 years represents approximately 18%. In the European SCT database, the number of patients aged > 65 years was <1% up to 2000 and 6.7% after 2000. This trend is the consequent to a growing clinical need caused to the progressive global aging of general population and to the increasing proportion of subjects with good performance status among elderly patients.

Fitness to transplantation is currently measured by the absence of the major comorbidities assessed by Sorror's Comorbidity Index score (HCT-CI). The score correlates with the outcome after transplant and provides clear indications on the intensity of the chemotherapy to be administered in pre-transplant phase in order to reduce Non Relapse Mortality (NRM).NRM is the mortality not due to the recovery of the disease; it can arise from three orders of complications: immunological (Graft versus Host Disease -GVHD-); infectious (opportunistic infections) and toxic (organ toxicity related to chemotherapy). The intensity of conditioning regimen is reduced consequently in presence of comorbidity and in the elderly patient, more frequently affected by comorbidities. But reducing the intensity of conditioning regimen also means significantly increasing the probability of relapse of haematological disease and therefore this reduction must be made on the basis of indexes of aging and comorbidity, as mentioned above (HCT-CI), in order to not overly reduce the curative potential of the transplant.This study aims to apply innovative markers of biological age for the evaluation of SCT patients. Biological age assessment is a rapidly expanding research area that has produced very promising results. Biological age is an index composed of molecular markers (such as DNA methylation of nucleated blood cells or the level of glycans associated with circulating proteins); it is strongly related to chronological age, but is capable of expressing the speed of aging of the single subject and consequently is able to highlight the risks for health associated with aging, with more emphasis than chronological age. The recent literature clearly indicates that DNA is also present in the non-cellular fraction, in the form of free DNA that it is largely contained in the compartment of nanovesicles. In particular, it is interesting to study if nanovesicles DNA can provide useful data regarding the epigenome and to verify how the epigenome is linked with the presence of exogenous DNA, that is the microbiome.This entity includes all the bacterial and viral species that coexist with every human, mostly located in the gastrointestinal tract, and which are increasingly determining to understand the pathogenesis of inflammatory and/or metabolic diseases, as well as the biological bases of aging. In this regard, the recent literature shows a close relationship between GVHD, viroma and intestinal microbiome.Epigenetics does not specifically deal with the modification of the sequence of the subject's DNA but with all the regulatory processes that influence gene expression. In particular, methylation is an epigenetic modification of DNA. Therefore, epigenetic studies differ from classical genetic studies in which the analysis of the exact DNA sequence of the subjects is carried out. In this protocol, the investigators will refer to the "study of DNA" as the study of its modifications in the methylation status and not in its sequence.

Primary objective of the study:

- Study of DNA in samples of patients undergoing allogeneic haematopoietic stem cell transplantation. In particular, DNA will be extracted from leukocytes and plasma extracellular nanovesicles. DNA will be assessed for the extent of methylation, which will be also in relationship with circulating exogenous DNA (i.e the microbiome).

Secondary objectives:

* Study of DNA in urine and faeces samples of the same subjects to describe further elements of the systemic microbiome - namely the urinary virome and the intestinal microbiome-.
* Correlation of circulating epigenome and systemic microbiome with clinical outcomes (overall survival, GVHD, incidence of infections) and comorbidity index (HCT-CI).

Exclusion criteria:

- Absence of signed informed consent.

No treatment is provided; patients will be treated and followed according to normal clinical practice and according to international guidelines.

The visits and evaluations are those of routine practice will not be modified. Samples of different biological materials will be taken at the start of recovery, at day -1, +1, and after 1, 3, 6, 9, 12 months after transplantation. After discharge, all patients will be followed as usual by the Day Hospital of the Transplant Unit of the Hematology Institute, where the prospective collection of samples at defined times will continue.

The primary objective of the study is descriptive. The evaluation of the main clinical variables is done with descriptive analysis (mean, median, range, etc.). Survival analysis will be performed according to Kaplan-Meier methodology for censored data. Regression analysis for censored data will be performed using Cox proportional risk models.

The DNA methylation is expressed in terms of continuous variables, as a percentage of methylation of the different analyzed gene loci. The analysis of methylation data will be performed through a pipeline of algorithms developed by the proponents. The viromic data are nominal variables (presence/absence of viral species).

The study is of exploratory nature and it is expected to enroll 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18.
* Patients with haematological disease undergoing allogeneic haematopoietic stem cell transplantation at "Seràgnoli" Hematology Institute, S. Orsola-Malpighi Hospital.
* Patients who consent to participate after signing written informed consent.

Exclusion Criteria:

- Absence of written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing allogeneic haematopoietic stem cell transplantation, as part of their normal pth of cure, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Study of DNA methylation | 24 months
  Study of DNA in samples of patients undergoing allogeneic haematopoietic stem cell transplantation. In particular, DNA will be extracted from leukocytes and plasma extracellular nanovesicles. DNA will be assessed for the extent of methylation, which will be also in relationship with circulating exogenous DNA (i.e the microbiome).

SECONDARY OUTCOMES:
Study of DNA for the determination of the systemic microbiome.. | 24 months
  Study of DNA in urine and faeces samples of the same subjects to describe further elements of the systemic microbiome - namely the urinary virome and the intestinal microbiome-.
Transplantation clinical outcomes. | 24 months
  Correlation of circulating epigenome and systemic microbiome with clinical outcomes (overall survival, GVHD, incidence of infections) and comorbidity index (HCT-CI).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bonifazi, MD, Principal Investigator — St. Orsola-Malpighi University Hospital, Bologna, Italy
Locations (1):
- St.Orsola-Malpighi University Hospital, Bologna, BO, Italy

REFERENCES:
- [Result] Bacalini MG, Gentilini D, Boattini A, Giampieri E, Pirazzini C, Giuliani C, Fontanesi E, Scurti M, Remondini D, Capri M, Cocchi G, Ghezzo A, Del Rio A, Luiselli D, Vitale G, Mari D, Castellani G, Fraga M, Di Blasio AM, Salvioli S, Franceschi C, Garagnani P. Identification of a DNA methylation signature in blood cells from persons with Down Syndrome. Aging (Albany NY). 2015 Feb;7(2):82-96. doi: 10.18632/aging.100715. PMID 25701644